CLINICAL TRIAL: NCT03819439
Title: Microbiome and Mycobiome Registry of Volunteers With and Without Autism Spectrum Disorder
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Mahmoiud A. Ghannoum, Director of Medical Mycology, University Hospitals Cleveland Medical Center
Other Study IDs: 03/18/29
Record Dates: First submitted 2019-01-15; First posted 2019-01-28 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; microbiome; mycobiome; bacteria; fungi
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: None Retained — stool samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Microbiome and Autism Questionnaire — The questionnaire will be administered to collect demographic data (i.e. sex, age, race, and ethnicity) of the volunteers. Additionally, it will ask for the volunteers to identify whether or not they have autism spectrum disorder and what other medical conditions they have and what medications (e.g. prescribed, over the counter, herbal; etc.) that they take.

SUMMARY:
Analyze, describe, and understand how the human gut microbiome (i.e. bacteriome and mycobiome) and Autism Spectrum Disorder (ASD) are related.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers > 2 years of age
* Able to list all medical conditions and medications when applicable.
* Have already donated a stool sample to BIOHM™.

Exclusion Criteria:

* Volunteers < 2 years of age

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Volunteers will or will not have a diagnosis of Autism Spectrum Disorder (ASD). Volunteers will be both local and national. There will be no limit to the number of volunteers who participate; however, we anticipate being able to enroll at least 50 volunteers within the first year.
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-07-23 (Actual)

PRIMARY OUTCOMES:
Characterize the microbiome [bacteria and fungal community] | 10 years
  Identifying relative abundance of individual bacterial and fungal members.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No